CLINICAL TRIAL: NCT01155076
Title: Effects of a Proprietary Ginseng, Cordyceps, and Pomegranate Supplement on Physical and Mental Function in Middle-aged Adults: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Effects of a Vitality Dietary Supplement on Physical and Mental Function in Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10-SUS-03-NU-01
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Health-related Quality of Life

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitality product (Experimental): Proprietary blend of ginseng, cordyceps, and pomegranate
  Interventions: Dietary Supplement: Vitality Product
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitality Product — Proprietary blend of ginseng, cordyceps, and pomegranate taken twice a day for 8 weeks
  Arms: Vitality product
Dietary Supplement: Placebo — Placebo taken twice a day for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effects of 8 weeks Vitality Product supplementation on physical and mental function in middle-aged adults

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40-70 years
* Signed Informed Consent
* BMI between 19 and 30 kg/m2
* Normotensive, defined as systolic blood pressure 90-140 mmHg and diastolic blood pressure 50-90 mmHg

Exclusion Criteria:

* Regular dietary supplement use and unwilling to discontinue use at least 1 month prior to enrollment in the study
* Self-reported chronic condition that may affect subject safety (e.g. diabetes, cardiovascular disease) or significantly impact product effectiveness (e.g. chronic fatigue)
* Pregnancy/suspected pregnancy, breastfeeding
* Antihypertensive medication use
* Allergies to any supplement ingredients
* Consumption of more than 600mg caffeine from any source per day
* Consumption of "energy drinks" (e.g. Red Bull, Monster) or any herbal supplement known to affect energy levels
* Known iron anemia
* Medically treated for insomnia
* Medically treated for depression
* Taking medications known to affect energy, e.g. thyroid medication
* Tobacco user
* Planned surgical procedure in next 2 months
* Participating in another clinical (medical or nutritional) study or likely to enroll in another medical or nutritional study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 8 weeks

SECONDARY OUTCOMES:
Medical Outcomes Study (MOS) Sexual Function questionnaire | 8 weeks
Adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John McGettigan, MD, Principal Investigator — Quality of Life Medical & Research Center, LLC
Locations (3):
- United States (3):
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Ridgeview Chaska Medical Plaza, Chaska, Minnesota
  - West Houston Clinical Research Services, Houston, Texas